CLINICAL TRIAL: NCT01281267
Title: Transplantation of Allograft Face or Facial Subunit for Treatment of Severe Facial Deformation
Brief Title: Face Transplantation for Treatment of Severe Facial Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bodhan Pomahac, Medical Director, Burn Center, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008P000550; W911QY09C0216 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Severe Facial Deformity
Keywords: facial transplantation; face transplantation; composite tissue allotransplantation; VCA; composite tissue allograft; facial allograft
MeSH Terms: interventions — Facial Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Face transplantation (Experimental)
  Interventions: Procedure: Facial Allograft Transplantation

INTERVENTIONS:
Procedure: Facial Allograft Transplantation — Facial allograft transplantation surgery is the transfer of face tissue from a deceased human donor to a patient with a severe facial deformity.
  Other Names: face transplantation; facial transplantation; composite facial allograft transplantation

SUMMARY:
Face transplantation surgery is the transfer of face tissue from a deceased human donor to a patient with a severe facial deformity. Face transplantation is an innovative reconstructive procedure that has the potential to significantly improve the lives of patients with severe facial injuries. The purpose of this study is to develop the best practices for facial transplantation that will improve the outcomes of future face transplant recipients.

DETAILED DESCRIPTION:
The United States Department of Defense (DoD) awarded Brigham and Women's Hospital (BWH) a research contract to fund 5 face transplantation surgeries.

The investigators are now actively seeking candidates for the procedure. The primary requirements to be considered as a candidate for face transplant surgery are: at least 18 years old; lost a major part of the face, such as the nose or the lips, or lost at least 25% of their facial tissue; and the facial injury cannot be treated acceptably by conventional reconstructive surgery. There are number of other factors that the investigators consider to determine who would be a suitable candidate.

From the time the investigators begin our search for a qualified face transplant recipient to the continuing care the investigators provide following surgery, a significant amount of time, expertise, and attentiveness is contributed toward making the procedure a progressive success. Below is an overview of what happens before, during and after a face transplant procedure.

Face transplant candidates go through an extensive screening process that is likely to last several months. This screening includes a psychiatric and social support evaluation and a series of imaging tests to help determine a patient's physical and mental readiness for the procedure. If, upon completion of the screening process, it is determined that a patient is a suitable candidate, the investigators will place the patient on a transplant waiting list. The investigators will then begin working to find a donor who matches the recipient's tissue requirements - e.g., similar age, right blood type. This search could take many months, and, if a suitable donor is not found within one year, the investigators will speak with the patient to determine whether they're willing to continue waiting. When a donor is found, the investigators will immediately inform the patient about when to arrive at the hospital for the operation. As the timing for this type of procedure is extremely important, patients are expected to be readily available.

The area most likely to be reconstructed in a face transplant is the central region of the face, which includes the nose and lips, as these facial structures are the most difficult to reconstruct with conventional plastic surgery techniques. In our most recent case, the face transplant included the entire nose; the soft tissues of the mid-face, including all its blood vessels, muscles, and nerves; and a significant portion of the mid-facial skeleton. Surgeons will then connect the facial graft blood vessels to the patient's blood vessels under a microscope to restore blood circulation before connecting nerves and other tissue, such as bone, cartilage and muscles, as needed.

While the face transplant is taking place, a separate, smaller surgery will also be performed. The investigators will take a skin sample (graft) from the arm of the donor and then attach the sample to the patient's chest or abdomen. The intent is to have the graft behave like the face transplant tissue, eventually becoming part of the patient's own skin. This is done so that later the investigators can take tiny samples (biopsies) of the new chest/abdomen tissue to look for signs of rejection, thereby minimizing the need to disturb the new face tissue after surgery.

Immediately after surgery, the face transplant recipient will be taken to the Intensive Care Unit (ICU) for observation. The patient will typically stay in the ICU for one or two days and then be moved to a private room. At this point, a physical therapist will help the patient regain as much facial movement as possible, and a psychiatrist will discuss any psychological concerns.

The patient will stay in the hospital until both the plastic surgery and medical transplant teams agree that it is safe for the patient to return home. This post-operative stay is anticipated to be approximately 7-14 days, but can vary due to a number of factors.

Following their discharge, face transplant patients will need to return to BWH for routine visits. These visits will include monitoring transplant drug levels (immune suppressants) through regular blood tests, imaging tests, assessing quality of life and checking for the return of sensation and movement to the face. The investigators will also periodically examine small tissue samples from the chest/abdomen graft under a microscope to look for any signs of rejection. These visits will typically take place on a weekly basis for the first three months and then at least once a month for the first year following surgery.

After the first year, it is expected that face transplant patients will need to visit the hospital less and less as time passes. However, patients should be prepared to make a lifetime commitment to immune suppressants to help prevent the rejection of the transplanted face tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Loss of a major part of the face, such as the nose or the lips, or at least 25% of the facial tissue.
* The facial defect cannot be restored with traditional reconstruction techniques.
* Signed written informed consent.
* Willing to complete psychological and social evaluations.
* Willing to take immunosuppressants - drugs that help prevent rejection of the transplant - for life.
* Willing to return for follow-up visits as determined by the treating physician and to comply with extensive post-transplant rehabilitation therapy.
* Willing to receive standard vaccinations prior to the transplant, such as influenza and hepatitis B.

Exclusion Criteria:

* Active malignancy.
* High risk of return of malignancy.
* History of persistent non-compliance.
* Findings of psychological evaluation that indicate inability to comply with physician's orders or mental instability.
* Any diagnosis that puts the subject at risk during the face transplant surgery.
* Absence of adequate donor sites for skin grafting in the event of transplant failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Outcomes of face transplantation. | Subjects will be followed for 18 months after face transplantation
  We will undertake an objective evaluation of the results of face transplantation in an 'outcome-oriented study'.

SECONDARY OUTCOMES:
Efficacy and optimization of the immune suppression protocol. | 18 months
  We will evaluate the risks of rejection or likelihood of tolerance induction by measuring specific parameters in the blood or tissue, including: Serum alloantibodies concentration, numbers/phenotype of specific T cell alloreactivity in the peripheral blood, phenotypic characterization of graft infiltrating cells and local gene expression of cells and cytokines.
Procedural outcomes of face transplantation | From subject recruitment to 18 months after transplantation
  We will optimize the screening, pre-operative, peri-operative and follow-up procedures of face transplantation.
Functional outcomes of face transplantation | Subjects will be followed for 18 months following face transplantation
  We will evaluate the return of facial sensory and motor function after face transplantation.
Psychosocial outcomes of face transplantation | Subjects will be followed up for 18 months following face transplantation
  We will evaluate the psychological and social outcomes of face transplantation by evaluating the subject's quality of life at various time points before and after transplantation.
Financial and economic aspects of face transplantation | Subjects will be followed for 18 months after face transplantation
  We will evaluate the cost-effectiveness of face transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Pomahac, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Pomahac B, Aflaki P. Composite tissue transplantation: a new era in transplantation surgery. Eplasty. 2010 Sep 15;10:e58. PMID 20862294
- [Background] Aflaki P, Nelson C, Balas B, Pomahac B. Simulated central face transplantation: age consideration in matching donors and recipients. J Plast Reconstr Aesthet Surg. 2010 Mar;63(3):e283-5. doi: 10.1016/j.bjps.2009.08.013. Epub 2009 Sep 13. No abstract available. PMID 19748842
- [Background] Pomahac B, Aflaki P, Nelson C, Balas B. Evaluation of appearance transfer and persistence in central face transplantation: a computer simulation analysis. J Plast Reconstr Aesthet Surg. 2010 May;63(5):733-8. doi: 10.1016/j.bjps.2009.01.078. Epub 2009 Apr 23. PMID 19398394
- [Background] Kiwanuka H, Bueno EM, Diaz-Siso JR, Sisk GC, Lehmann LS, Pomahac B. Evolution of ethical debate on face transplantation. Plast Reconstr Surg. 2013 Dec;132(6):1558-1568. doi: 10.1097/PRS.0b013e3182a97e2b. PMID 24281583
- [Background] Lamparello BM, Bueno EM, Diaz-Siso JR, Sisk GC, Pomahac B. Face time: educating face transplant candidates. Eplasty. 2013 Jul 4;13:e36. Print 2013. PMID 23861990
- [Result] Soga S, Ersoy H, Mitsouras D, Schultz K, Whitmore AG, Powers SL, Steigner ML, Signorelli J, Prior RF, Rybicki FJ, Pomahac B. Surgical planning for composite tissue allotransplantation of the face using 320-detector row computed tomography. J Comput Assist Tomogr. 2010 Sep-Oct;34(5):766-9. doi: 10.1097/RCT.0b013e3181e9c133. PMID 20861783
- [Result] Pomahac B, Pribaz J, Eriksson E, Annino D, Caterson S, Sampson C, Chun Y, Orgill D, Nowinski D, Tullius SG. Restoration of facial form and function after severe disfigurement from burn injury by a composite facial allograft. Am J Transplant. 2011 Feb;11(2):386-93. doi: 10.1111/j.1600-6143.2010.03368.x. Epub 2011 Jan 7. PMID 21214855
- [Result] Edrich T, Pomahac B, Lu JT, Couper GS, Gerner P. Perioperative management of partial face transplantation involving a heparin antibody-positive donor. J Clin Anesth. 2011 Jun;23(4):318-21. doi: 10.1016/j.jclinane.2010.07.004. PMID 21663819
- [Result] Pomahac B, Nowinski D, Diaz-Siso JR, Bueno EM, Talbot SG, Sinha I, Westvik TS, Vyas R, Singhal D. Face transplantation. Curr Probl Surg. 2011 May;48(5):293-357. doi: 10.1067/j.cpsurg.2011.01.003. No abstract available. PMID 21463717
- [Result] Pomahac B, Lengele B, Ridgway EB, Matros E, Andrews BT, Cooper JS, Kutz R, Pribaz JJ. Vascular considerations in composite midfacial allotransplantation. Plast Reconstr Surg. 2010 Feb;125(2):517-522. doi: 10.1097/PRS.0b013e3181c82e6f. PMID 19910848
- [Result] Saavedra AP, Bueno EM, Granter SR, Pomahac B. Transmission of donor-specific skin condition from donor to recipient of facial allograft. Am J Transplant. 2011 Jun;11(6):1340. doi: 10.1111/j.1600-6143.2011.03596.x. No abstract available. PMID 21645261
- [Result] Kumamaru KK, Sisk GC, Mitsouras D, Schultz K, Steigner ML, George E, Enterline DS, Bueno EM, Pomahac B, Rybicki FJ. Vascular communications between donor and recipient tissues after successful full face transplantation. Am J Transplant. 2014 Mar;14(3):711-9. doi: 10.1111/ajt.12608. Epub 2014 Feb 6. PMID 24502329
- [Result] Lian CG, Bueno EM, Granter SR, Laga AC, Saavedra AP, Lin WM, Susa JS, Zhan Q, Chandraker AK, Tullius SG, Pomahac B, Murphy GF. Biomarker evaluation of face transplant rejection: association of donor T cells with target cell injury. Mod Pathol. 2014 Jun;27(6):788-99. doi: 10.1038/modpathol.2013.249. Epub 2014 Jan 17. PMID 24434898
- [Result] Sinha I, Pomahac B. Split rejection in vascularized composite allotransplantation. Eplasty. 2013 Oct 8;13:e53. PMID 24244785
- [Result] Schultz K, George E, Mullen KM, Steigner ML, Mitsouras D, Bueno EM, Pomahac B, Rybicki FJ, Kumamaru KK. Reduced radiation exposure for face transplant surgical planning computed tomography angiography. PLoS One. 2013 Apr 26;8(4):e63079. doi: 10.1371/journal.pone.0063079. Print 2013. PMID 23638180
- [Result] Pomahac B, Bueno EM, Sisk GC, Pribaz JJ. Current principles of facial allotransplantation: the Brigham and Women's Hospital Experience. Plast Reconstr Surg. 2013 May;131(5):1069-1076. doi: 10.1097/PRS.0b013e3182865cd3. PMID 23629089
- [Derived] Win TS, Crisler WJ, Dyring-Andersen B, Lopdrup R, Teague JE, Zhan Q, Barrera V, Ho Sui S, Tasigiorgos S, Murakami N, Chandraker A, Tullius SG, Pomahac B, Riella LV, Clark RA. Immunoregulatory and lipid presentation pathways are upregulated in human face transplant rejection. J Clin Invest. 2021 Apr 15;131(8):e135166. doi: 10.1172/JCI135166. PMID 33667197
- [Derived] Aycart MA, Alhefzi M, Sharma G, Krezdorn N, Bueno EM, Talbot SG, Carty MJ, Tullius SG, Pomahac B. Outcomes of Solid Organ Transplants After Simultaneous Solid Organ and Vascularized Composite Allograft Procurements: A Nationwide Analysis. Transplantation. 2017 Jun;101(6):1381-1386. doi: 10.1097/TP.0000000000001262. PMID 27140518
- [Derived] Borges TJ, O'Malley JT, Wo L, Murakami N, Smith B, Azzi J, Tripathi S, Lane JD, Bueno EM, Clark RA, Tullius SG, Chandraker A, Lian CG, Murphy GF, Strom TB, Pomahac B, Najafian N, Riella LV. Codominant Role of Interferon-gamma- and Interleukin-17-Producing T Cells During Rejection in Full Facial Transplant Recipients. Am J Transplant. 2016 Jul;16(7):2158-71. doi: 10.1111/ajt.13705. Epub 2016 Apr 7. PMID 26749226
- [Derived] Soga S, Pomahac B, Mitsouras D, Kumamaru K, Powers SL, Prior RF, Signorelli J, Bueno EM, Steigner ML, Rybicki FJ. Preoperative vascular mapping for facial allotransplantation: four-dimensional computed tomographic angiography versus magnetic resonance angiography. Plast Reconstr Surg. 2011 Oct;128(4):883-891. doi: 10.1097/PRS.0b013e3182268b43. PMID 21921764
- See also: Study's official webpage — https://www.brighamandwomens.org/surgery/plastic-surgery/restorative-surgery/face-transplant-surgery